CLINICAL TRIAL: NCT06667596
Title: The Effect of Anaesthesia Technique on Preoperative Fear of Death and Anxiety in Upper Extremity Surgery Patients
Brief Title: The Effect of Anaesthesia Technique on Anxiety in Upper Extremity Surgery Patients
Status: Withdrawn | Type: Observational
Why Stopped: The ethics committee did not approve it.
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Emine OZCAN, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: EK3604
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Preoperative Anxiety
Keywords: Preoperative anxiety; Upper extremity surgery; Peripheric nerve block; Regional Anesthesia; General Anesthesia; Anesthesia Anxiety; Surgery Anxiety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anxiety: Patients aged 18-65 years, ASA-I-II-III, oriented and cooperative, who agreed to participate in the survey, undergoing upper extremity surgery under regional or general anesthesia.

SUMMARY:
This prospective, cross-sectional study aims to investigate the impact of planned anesthesia technique (general or regional anesthesia) and patients' previous anesthesia experience on preoperative anxiety in patients undergoing upper extremity surgery. The secondary objective is to identify the reasons for patients' anxiety related to anesthesia and surgery. Preoperative anxiety can lead to emotional, psychiatric, and physical problems, and is associated with increased autonomic fluctuations, anesthetic demand, postoperative nausea and vomiting, pain, prolonged recovery time, and hospitalization. The study will enroll 400 volunteers undergoing upper extremity surgery at Başakşehir Çam and Sakura City Hospital. Demographic information, surgical details, previous surgical and psychiatric history, substance abuse, and information about anesthesia will be collected. The Amsterdam Preoperative Anxiety and Information Form (APAIS) will be used to assess anxiety and desire for information, while the State-Trait Anxiety Inventory (STAI) will evaluate state and trait anxiety. Patients with an APAIS-A score ≥13 will be considered anxious, and those with an APAIS-B score ≥4 will be considered information-seeking. STAI scores will be interpreted based on percentile ranks and average score levels. The study aims to identify approaches to reduce preoperative anesthesia and surgery-related anxiety. SPSS Survey Analysis methods will be used for statistical analysis. The study duration is 12 months, from November 2024 to November 2025. Inclusion criteria are consenting patients aged 18-65 years, ASA I-III, undergoing upper extremity surgery under general or regional anesthesia, who are oriented and cooperative. Exclusion criteria include lack of consent, inappropriate age, ASA IV-V, non-upper extremity surgery, and inability to orient and cooperate.

DETAILED DESCRIPTION:
RESEARCH PROTOCOL

1. The full name of the study:

   The Effect of Anaesthesia Technique on Preoperative Fear of Death and Anxiety in Upper Extremity Surgery Patients
2. Purpose and importance of the research (primary purpose, secondary purposes, if any):

   Preoperative anxiety is one of the most important problems for patients. Because it causes emotional and psychiatric problems as well as physical problems. To help patients, it is very important to identify the patient's current anxiety. Our primary aim in this study is to investigate how the planned anesthesia technique (general anesthesia or regional anesthesia) and the patients' previous anesthesia experience affect the patient's anxiety in patients undergoing upper extremity surgery (shoulder, arm, wrist, hand). Our secondary aim is to reveal the reasons for patients' anxiety about anesthesia and surgery.
3. Expected benefits and risks of the research:

   Preoperative anxiety is very important as it has the potential to affect all aspects of anesthesia, including preoperative assessment, induction of anesthesia, perioperative and recovery periods. The exact etiology of anxiety may be related to anesthesia, surgery and many other causes. Perioperative anxiety is known to be associated with increased autonomic fluctuations and anesthetic demand, increased incidence of nausea and vomiting, and increased pain in the postoperative period. As a consequence of these complications, prolonged recovery time and hospitalization have been reported. In patients undergoing upper extremity surgery (shoulder, arm, wrist, hand), the anxious conditions caused by being close to the surgical site and team may vary according to the application of general anesthesia or regional anesthesia technique. With this study, we seek to answer the question 'what approaches should we develop to reduce the level of anxiety related to preoperative anesthesia and surgery in patients? Therefore, identifying and preventing patients' current anxiety to help patients are the benefits we expect. Since it will be a question and answer study with face-to-face interviews in the preoperative period in patients who will undergo upper extremity surgery, which is routinely performed in our hospital, there is no risk.
4. Type, scope and design of the planned study:

   Prospective, Cross-Sectional In our study, patients who will undergo upper extremity surgery will be asked whether they want to participate in the preoperative period, face-to-face anesthesia and surgery-induced anxiety and its causes, we plan to conduct a survey consisting of several questions to determine the effect of anesthesia technique on their anxiety and whether they want to participate in it. After obtaining informed consent for the survey from the volunteer patients in the preoperative patient preparation room, demographic information and questions in the scales (Amsterdam preoperative anxiety and information form (APAIS), STAI FORM TX-1 and TX-2) will be asked face to face. The answers received from the patients will be calculated according to the scoring system specified in the scales and anxiety levels will be determined. The aim of our study is to determine the effects of anesthesia technique on anxiety and fear of death in patients undergoing upper extremity surgery. To find ways to reduce anxiety in terms of anesthesia for patients.
5. The number of patients and volunteers to be included in the study, their qualifications and rationale for selection (age ranges, gender, etc.).

   Volunteers will be selected among the patients who will undergo upper extremity surgery (shoulder, arm, wrist, hand) in the Orthopedics and Hand Surgery Clinics of Başakşehir Çam and Sakura City Hospital after ethics committee approval is obtained. The statistical sample size calculation was found to be 400 patients as a result of the statistical sample size calculation considering a 5% margin of error at 95% confidence interval.
6. Parameters to be checked (must be written individually and clearly) Age, gender, education and marital status of the patients, what kind of surgery they will have, whether they know their surgeon, whether they have been informed about the surgery and its risks, whether they have had surgery before, if so, what is their experience, have they received psychiatric treatment in the past and are they still receiving psychiatric treatment? Is there any alcohol or substance abuse? Did he/she have an interview with the anesthesiologist before the operation? Has he/she been informed about anesthesia? Which anesthesia technique will be used for the operation? Has he/she been informed about this? This information will be asked and recorded. Amsterdam Preoperative Anxiety and Information Form will be used for anxiety and request for information and the results will be recorded.

   AMSTERDAM PREOPERATIVE ANXIETY AND INFORMATION FORM: The APAIS form includes 6 statements measuring anxiety and desire for information. Patients will be asked to give a value between 1-5 to 4 statements measuring anxiety (1, 2, 4 and 5.) and 2 statements measuring desire for information (3 and 6). The sum of the values given to the statements measuring anxiety constitutes the APAIS-A anxiety score, and the sum of the values given to the statements measuring the desire for information constitutes the APAIS-B desire for information score. Patients with an APAIS-A anxiety score of 13 and above will be considered as 'feeling anxious' and patients with an APAIS-B information seeking score of 4 and above will be considered as 'seeking information'. Is the patient's surgery induced? State and Trait Anxiety Scale Scoring will be used to assess whether the patient is personally anxious.

   STAI FORM TX - I and STAI FORM TX-2 ( STATE AND TRAIT ANXIETY SCALE SCORING ) : If more than three answers are not given to a statement, the completed form is considered invalid and not scored. Response options collected in four classes in the state anxiety scale, (1) Not at all, (2) A little, (3) A lot and (4) Completely The options in the Trait Anxiety Scale are (1) Almost never, (2) Sometimes, (3) Very often and (4) Almost always.

   There are two types of expressions in scales. We can call them 1) direct or straight statements and 2) reversed statements. Direct statements express negative emotions, while reversed statements express positive emotions. When scoring these second type of statements, those with a score of 1 turn into 4 and those with a score of 4 turn into 1. In direct statements, answers with a value of 4 indicate that anxiety is high. In inverted statements, answers with a value of 1 indicate high anxiety and answers with a value of 4 indicate low anxiety. The expression "I am restless" can be shown as an example of direct statements and the expression "I feel calm" can be shown as an example of inverted statements. In this case, if an option with a weight of 4 is selected for the expression "I feel restless" and an option with a weight of 1 is selected for the expression "I feel calm", these answers reflect high anxiety.

   There are ten inverted statements in the state anxiety scale. These are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20.

   In the trait anxiety scale, the number of inverted statements is seven and these are items 21, 26, 27, 30, 33, 36 and 39.

   Two separate keys are prepared for each of the direct and reverse statements. Thus, the total weights of the direct statements are calculated with one key and the total weights of the reversed statements are calculated with the second key. The total weighted score for the direct statements is subtracted from the total weighted score for the reverse statements. A predetermined and unchanging value is added to this number.

   This constant value for the state anxiety scale is 50, For the trait anxiety scale, it is 35. The last value obtained is the anxiety score of the individual. INTERPRETATION OF SCORES The scores obtained from both scales theoretically range between 20 and 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety. The same is true when the scores are interpreted in percentile order. In other words, a low percentile rank (1, 5, 10) indicates a low level of anxiety. The average score level determined in the applications varied between 36 and 41.

   The anxiety levels of the patients will be determined according to the scoring system in these scales.
7. Where and by whom to look at the parameters

   Başakşehir Çam and Sakura will be cared for by Specialist Dr. Emine Özcan and Specialist Dr. Abdurrahman Engin Baydemir at the City Hospital.
8. Which of the parameters to be used in the study are routine for that disease group and which are specific to the study,

   APAIS (Amsterdam Preoperative Anxiety and Information Form) and STAI FORM TX-1 (State Anxiety Scale) and STAI FORM TX-2 (Trait Anxiety Scale) are the scales used for Anxiety.
9. Anticipated duration of work, start and end dates,

12 months 04.11.2024 - 01.11.2025

10. Inclusion, exclusion and withdrawal criteria, Inclusion criteria;

* Consenting patients,
* 18-65 years old,
* ASA-I-II-III
* He will undergo upper extremity (shoulder, arm, wrist, hand) surgery,
* He will receive General or Regional Anesthesia,
* Oriented and cooperative patients, Exclusion criteria;
* Patients without consent,
* Not in the appropriate age range,
* Patients with ASA-IV-V,
* Those who will not undergo upper extremity surgery,
* Patients who cannot orient and cooperate

  11. Criteria for terminating the research, Reaching a predetermined number of patients or time limitation.

  12. In the evaluation of the data to be obtained as a result of the research The statistical methods to be used should be explained, SPSS (Statistical Package for the Social Sciences) Survey Analysis methods will be used

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients,
* 18-65 years old,
* ASA-I-II-III
* They will undergo upper extremity (shoulder, arm, wrist, hand) surgery,
* They will receive General or Regional Anesthesia,
* Oriented and cooperative patients,

Exclusion Criteria:

* Patients without consent,
* Not in the appropriate age range,
* Patients with ASA-IV-V,
* Those who will not undergo upper extremity surgery,
* Patients who cannot orient and cooperate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be selected among the patients who will undergo upper extremity surgery (shoulder, arm, wrist, hand) in the Orthopedics and Hand Surgery Clinics of Başakşehir Çam and Sakura City Hospital after ethics committee approval is obtained. The statistical sample size calculation was found to be 400 patients as a result of the statistical sample size calculation considering a 5% margin of error at 95% confidence interval.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2026-12-02 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
APAIS (The Amsterdam Preoperative Anxiety and Information Scale) | November 2024- June 2025
  The Amsterdam Preoperative Anxiety and Information Scale The APAIS form includes 6 statements measuring anxiety and desire for information. Patients will be asked to give a value between 1-5 to 4 statements measuring anxiety (1, 2, 4 and 5.) and 2 statements measuring desire for information (3 and 6). The sum of the values given to the statements measuring anxiety constitutes the APAIS-A anxiety score, and the sum of the values given to the statements measuring the desire for information constitutes the APAIS-B desire for information score. Patients with an APAIS-A anxiety score of 13 and above will be considered 'anxious' and patients with an APAIS-B information seeking score of 4 and above will be considered 'seeking information'.

SECONDARY OUTCOMES:
STAI-TX-1( State Anxiety Scale) and STA-TX-2 (Trait Anxiety Scale) | November 2024- June 2025
  Application of State-Trait Anxiety Scale (STAI-TX) INTERPRETATION OF SCORES The scores obtained from both scales theoretically range between 20 and 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety. The same is true when the scores are interpreted in percentile order. In other words, a low percentile rank (1, 5, 10) indicates a low level of anxiety. The average score level determined in the applications varied between 36 and 41.
  The anxiety levels of the patients will be determined according to the scoring system in these scales.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Ozcan, Principal Investigator, Principal Investigator — Başakşehir Çam ve Sakura Şehir Hastanesi
Locations (1):
- Başakşehir Çam ve Sakura Şehir Hastanesi, Istanbul, Başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh J, Lee W, Ki S, Suh J, Hwang S, Lee J. Assessment of Preoperative Anxiety and Influencing Factors in Patients Undergoing Elective Surgery: An Observational Cross-Sectional Study. Medicina (Kaunas). 2024 Feb 27;60(3):403. doi: 10.3390/medicina60030403. PMID 38541129
- [Background] Salzmann S, Rienmuller S, Kampmann S, Euteneuer F, Rusch D. Preoperative anxiety and its association with patients' desire for support - an observational study in adults. BMC Anesthesiol. 2021 May 17;21(1):149. doi: 10.1186/s12871-021-01361-2. PMID 34000986
- [Background] Eberhart L, Aust H, Schuster M, Sturm T, Gehling M, Euteneuer F, Rusch D. Preoperative anxiety in adults - a cross-sectional study on specific fears and risk factors. BMC Psychiatry. 2020 Mar 30;20(1):140. doi: 10.1186/s12888-020-02552-w. PMID 32228525
- [Background] Sertcakacilar G, Yildiz GO, Bayram B, Pektas Y, Cukurova Z, Hergunsel GO. Comparing Preoperative Anxiety Effects of Brachial Plexus Block and General Anesthesia for Orthopedic Upper-Extremity Surgery: A Randomized, Controlled Trial. Medicina (Kaunas). 2022 Sep 16;58(9):1296. doi: 10.3390/medicina58091296. PMID 36143973
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/